CLINICAL TRIAL: NCT04921176
Title: Evaluating Quality of Life of AF Patients Following a Bleed
Acronym: EQUAL-AF
Status: Completed | Type: Observational
Sponsor: Swansea University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 279646
Record Dates: First submitted 2021-01-27; First posted 2021-06-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
Keywords: Quality of Life; Bleed events; Patient Reported Outcome Measure; Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
EQUAL-AF is an observational feasibility study which will determine if there is a long-term effect of bleeding for patients diagnosed with AF, who are taking anticoagulants. The investigators will use three validated questionnaires/PROMs (AFEQT, EQ5D-3L, and PACT-Q) to gather data from a patient perspective. Patients will complete all questionnaires no more than 4 weeks following a bleed and a second time 3 months later. As this study tests feasibility, progression criteria will apply. The primary objective is to assess recruitment success to ensure that the patient population is accessible and willing to engage with the research team. Additionally, the investigators will look to identify the need for a specific bleeding PROM which will assess long-term quality of life impact for patients experiencing bleeds while anticoagulated.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (>= 18 years old)
* Patients who can understand all study information and literature to provide fully informed consent
* Atrial fibrillation (AF) as the primary diagnosis
* Having a major or minor bleed up to a maximum of 30 days prior to point of enrolment
* Receiving oral anticoagulation therapy for AF

Exclusion Criteria:

* Pregnant women
* Patients with active cancer
* Patients unable to consent for themselves
* Patient on concomitant antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18) who have AF are actively prescribed oral anticoagulant therapies (OATs) and have recently experienced bleeds, up to a maximum of 4 weeks prior to enrolment. No upper age limit will be applied, but patients must match all other inclusion/exclusion criteria. Patients will be selected from the Swansea area only, who attend/have attended either anticoagulation clinics within the Swansea City Health Cluster, Morriston emergency department or have been admitted to wards at Morriston Hospital due to a bleed.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Test the feasibility of identifying and recruiting patients with both minor and major bleeds as a result of anticoagulant treatment for AF associated events | Following 6 months recruitment window
  Recruitment of a minimum of 50 eligible patients onto the study
Patient quality of life in both primary and secondary care settings as measured by EQ-5D-5L score | Within 4 weeks following bleed
  Patient quality of life in both primary and secondary care settings as measured by EQ-5D-
Patient quality of life in both primary and secondary care settings as measured by EQ-5D-5L score | 3 months following first completion of study survey
  Patient quality of life in both primary and secondary care settings as measured by EQ-5D-
Patient quality of life in both primary and secondary care settings as measured by Atrial Fibrillation Effect of Quality of Life score (AFEQT) | Within 4 weeks following bleed
  Patient quality of life in both primary and secondary care settings as measured by Atrial
Patient quality of life in both primary and secondary care settings as measured by Atrial Fibrillation Effect of Quality of Life score (AFEQT) | 3 months following first completion of study survey
  Patient quality of life in both primary and secondary care settings as measured by Atrial
Patient quality of life in both primary and secondary care settings as measured by Perception of Anticoagulant Treatment Questionnaire (PACT-Q) | Within 4 weeks following bleed
  Patient quality of life in both primary and secondary care settings as measured by
Patient quality of life in both primary and secondary care settings as measured by Perception of Anticoagulant Treatment Questionnaire (PACT-Q) | 3 months following first completion of study survey
  Patient quality of life in both primary and secondary care settings as measured by

SECONDARY OUTCOMES:
Observe differences in QoL by type of bleed as measured by clinical classification of minor and major bleeds using BARC scale. | One data point at 4 weeks using the validated questionnaires and a follow-up at 3 months for each patient.
  A small number of additional relevant questions will be asked of the patient, regarding when the bleed occurred, the nature of the bleed and their current treatment.
Identifying the treatment received and the nature of the bleed experienced by capturing type of anticoagulant combined with bleed details from each participant. | One data point at 4 weeks using the validated questionnaires and a follow-up at 3 months for each patient.
  Identifying the treatment received and the nature of the bleed experienced by capturing
Insight into issues experienced with bleeding from participant perspective as measured by structured qualitative interviews. | Following completion of both 4 week and 3 month timepoint.
  Insight into issues experienced with bleeding from participant perspective as measured by structured qualitative interviews.
Appropriateness of three chosen PROMs (EQ5D, AFEQT and PACT-Q, part 2) in capturing QoL data for patients who have experienced a bleed while anticoagulated as measured by responses to suitability questions within the participant survey. | One data point at 4 weeks using the validated questionnaires and a follow-up at 3 months for each patient.
  Additional questions to evaluate appropriateness of chosen PROMs in capturing Quality of Life issues for patients diagnosed with AF who are anticoagulated

CONTACTS AND LOCATIONS:
Overall Officials: Hayley Hutchings, Principal Investigator — Swansea University
Locations (3):
- United Kingdom (3):
  - Arrhythmia Alliance, Oxford, England
  - Morriston Hospital, Swansea, West Glamorgan
  - Swansea City GP Cluster, Swansea, West Glamorgan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Liu GJ, Wang YF, Chen PY, Chang W, Tu ML, Chang LY, Cheng P, Luo J. The efficacy and safety of novel oral anticoagulants for the preventive treatment in atrial fibrillation patients: a systematic review and meta-analysis. Drug Deliv. 2014 Sep;21(6):436-52. doi: 10.3109/10717544.2013.873500. Epub 2014 Jan 8. PMID 24400656
- [Background] Patel NJ, Atti V, Mitrani RD, Viles-Gonzalez JF, Goldberger JJ. Global rising trends of atrial fibrillation: a major public health concern. Heart. 2018 Dec;104(24):1989-1990. doi: 10.1136/heartjnl-2018-313350. Epub 2018 Jun 15. No abstract available. PMID 29907645
- [Background] Darby-Stewart A, Dachs R, Graber MA. Rivaroxaban vs. warfarin for stroke prevention in patients with nonvalvular atrial fibrillation. Am Fam Physician. 2012 Mar 15;85(6):577-86. PMID 22534269
- [Background] Chugh SS, Havmoeller R, Narayanan K, Singh D, Rienstra M, Benjamin EJ, Gillum RF, Kim YH, McAnulty JH Jr, Zheng ZJ, Forouzanfar MH, Naghavi M, Mensah GA, Ezzati M, Murray CJ. Worldwide epidemiology of atrial fibrillation: a Global Burden of Disease 2010 Study. Circulation. 2014 Feb 25;129(8):837-47. doi: 10.1161/CIRCULATIONAHA.113.005119. Epub 2013 Dec 17. PMID 24345399
- [Background] Li X, Tse VC, Au-Doung LW, Wong ICK, Chan EW. The impact of ischaemic stroke on atrial fibrillation-related healthcare cost: a systematic review. Europace. 2017 Jun 1;19(6):937-947. doi: 10.1093/europace/euw093. PMID 27209573
- [Background] Lane DA, Skjoth F, Lip GYH, Larsen TB, Kotecha D. Temporal Trends in Incidence, Prevalence, and Mortality of Atrial Fibrillation in Primary Care. J Am Heart Assoc. 2017 Apr 28;6(5):e005155. doi: 10.1161/JAHA.116.005155. PMID 28455344
- [Background] Hansen PW, Sehested TSG, Fosbol EL, Torp-Pedersen C, Kober L, Andersson C, Gislason GH. Trends in warfarin use and its associations with thromboembolic and bleeding rates in a population with atrial fibrillation between 1996 and 2011. PLoS One. 2018 Mar 16;13(3):e0194295. doi: 10.1371/journal.pone.0194295. eCollection 2018. PMID 29547673
- [Background] Kannel WB, Wolf PA, Benjamin EJ, Levy D. Prevalence, incidence, prognosis, and predisposing conditions for atrial fibrillation: population-based estimates. Am J Cardiol. 1998 Oct 16;82(8A):2N-9N. doi: 10.1016/s0002-9149(98)00583-9. PMID 9809895
- [Background] Barra S, Fynn S. Untreated atrial fibrillation in the United Kingdom: Understanding the barriers and treatment options. J Saudi Heart Assoc. 2015 Jan;27(1):31-43. doi: 10.1016/j.jsha.2014.08.002. Epub 2014 Sep 3. PMID 25544820
- [Background] Montbleau KE, King D, Henault L, Magnani JW. Health literacy, health-related quality of life, and atrial fbrillation. Cogent Med. 2017;4:1412121. doi: 10.1080/2331205X.2017.1412121. Epub 2017 Dec 11. PMID 29276719
- [Background] Thrall G, Lane D, Carroll D, Lip GY. Quality of life in patients with atrial fibrillation: a systematic review. Am J Med. 2006 May;119(5):448.e1-19. doi: 10.1016/j.amjmed.2005.10.057. PMID 16651058
- [Background] Spertus J, Dorian P, Bubien R, Lewis S, Godejohn D, Reynolds MR, Lakkireddy DR, Wimmer AP, Bhandari A, Burk C. Development and validation of the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire in patients with atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):15-25. doi: 10.1161/CIRCEP.110.958033. Epub 2010 Dec 15. PMID 21160035
- [Background] Hagens VE, Ranchor AV, Van Sonderen E, Bosker HA, Kamp O, Tijssen JG, Kingma JH, Crijns HJ, Van Gelder IC; RACE Study Group. Effect of rate or rhythm control on quality of life in persistent atrial fibrillation. Results from the Rate Control Versus Electrical Cardioversion (RACE) Study. J Am Coll Cardiol. 2004 Jan 21;43(2):241-7. doi: 10.1016/j.jacc.2003.08.037. PMID 14736444
- [Background] Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Guyton RA, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Wann LS, Curtis AB, Ellenbogen KA, Estes NA 3rd, Ezekowitz MD, Jackman WM, January CT, Lowe JE, Page RL, Slotwiner DJ, Stevenson WG, Tracy CM, Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Le Heuzey JY, Kay GN, Olsson SB, Prystowsky EN, Tamargo JL, Wann S. Management of patients with atrial fibrillation (compilation of 2006 ACCF/AHA/ESC and 2011 ACCF/AHA/HRS recommendations): a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 May 7;61(18):1935-44. doi: 10.1016/j.jacc.2013.02.001. Epub 2013 Apr 1. No abstract available. PMID 23558044
- [Background] January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC Jr, Ellinor PT, Ezekowitz MD, Field ME, Furie KL, Heidenreich PA, Murray KT, Shea JB, Tracy CM, Yancy CW. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019 Jul 9;140(2):e125-e151. doi: 10.1161/CIR.0000000000000665. Epub 2019 Jan 28. No abstract available. PMID 30686041
- [Background] Xu J, Luc JG, Phan K. Atrial fibrillation: review of current treatment strategies. J Thorac Dis. 2016 Sep;8(9):E886-E900. doi: 10.21037/jtd.2016.09.13. PMID 27747025
- [Background] Wallis CJD, Juvet T, Lee Y, Matta R, Herschorn S, Kodama R, Kulkarni GS, Satkunasivam R, Geerts W, McLeod A, Narod SA, Nam RK. Association Between Use of Antithrombotic Medication and Hematuria-Related Complications. JAMA. 2017 Oct 3;318(13):1260-1271. doi: 10.1001/jama.2017.13890. PMID 28973248
- [Background] Gorman EW, Perkel D, Dennis D, Yates J, Heidel RE, Wortham D. Validation Of The HAS-BLED Tool In Atrial Fibrillation Patients Receiving Rivaroxaban. J Atr Fibrillation. 2016 Aug 31;9(2):1461. doi: 10.4022/jafib.1461. eCollection 2016 Aug-Sep. PMID 27909541
- [Background] Dar T, Yarlagadda B, Vacek J, Dawn B, Lakkireddy D. Management of Stroke risk in atrial fibrillation patients with bleeding on Oral Anticoagulation Therapy-Role of Left Atrial Appendage Closure, Octreotide and more. J Atr Fibrillation. 2017 Dec 31;10(4):1729. doi: 10.4022/jafib.1729. eCollection 2017 Dec. PMID 29487685
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Res LCS, Lubberts B, Shah SH, DiGiovanni CW. Health-related quality of life after adverse bleeding events associated with antithrombotic drug therapy - A systematic review. Hellenic J Cardiol. 2019 Jan-Feb;60(1):3-10. doi: 10.1016/j.hjc.2018.06.012. Epub 2018 Jul 24. PMID 29908761
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Badia X, Arribas F, Ormaetxe JM, Peinado R, de Los Terreros MS. Development of a questionnaire to measure health-related quality of life (HRQoL) in patients with atrial fibrillation (AF-QoL). Health Qual Life Outcomes. 2007 Jul 4;5:37. doi: 10.1186/1477-7525-5-37. PMID 17610734
- [Background] Bae JM. Value-based medicine: concepts and application. Epidemiol Health. 2015 Mar 4;37:e2015014. doi: 10.4178/epih/e2015014. eCollection 2015. PMID 25773441
- [Background] Riva S, Pravettoni G. Value-Based Model: A New Perspective in Medical Decision-making. Front Public Health. 2016 Jun 13;4:118. doi: 10.3389/fpubh.2016.00118. eCollection 2016. No abstract available. PMID 27379224
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Rodeghiero F, Tosetto A, Abshire T, Arnold DM, Coller B, James P, Neunert C, Lillicrap D; ISTH/SSC joint VWF and Perinatal/Pediatric Hemostasis Subcommittees Working Group. ISTH/SSC bleeding assessment tool: a standardized questionnaire and a proposal for a new bleeding score for inherited bleeding disorders. J Thromb Haemost. 2010 Sep;8(9):2063-5. doi: 10.1111/j.1538-7836.2010.03975.x. No abstract available. PMID 20626619
- [Background] Buchholz I, Janssen MF, Kohlmann T, Feng YS. A Systematic Review of Studies Comparing the Measurement Properties of the Three-Level and Five-Level Versions of the EQ-5D. Pharmacoeconomics. 2018 Jun;36(6):645-661. doi: 10.1007/s40273-018-0642-5. PMID 29572719
- [Background] De Caterina R, Bruggenjurgen B, Darius H, Kohler S, Lucerna M, Pecen L, Renda G, Schilling RJ, Schliephacke T, Zamorano JL, Le Heuzey JY, Kirchhof P. Quality of life and patient satisfaction in patients with atrial fibrillation on stable vitamin K antagonist treatment or switched to a non-vitamin K antagonist oral anticoagulant during a 1-year follow-up: A PREFER in AF Registry substudy. Arch Cardiovasc Dis. 2018 Feb;111(2):74-84. doi: 10.1016/j.acvd.2017.04.007. Epub 2017 Sep 21. PMID 28942115
- [Derived] Hutchings HA, Lanyon KJ, Holland G, Alikhan R, Jenkins R, Laing H, Hughes A, Lobban T, Pollock K, Tod D, Lister S. Can we collect health-related quality of life information from anticoagulated atrial fibrillation participants who have recently experienced a bleed? An observational feasibility study in primary and secondary care in Wales and through a UK online forum. BMJ Open. 2023 Oct 6;13(10):e075335. doi: 10.1136/bmjopen-2023-075335. PMID 37802619
- [Derived] Hutchings HA, Lanyon K, Lister S, Alikhan R, Halcox J, Holland G, Hughes A, Jenkins R, Laing H, Lobban T, Owen D, Pollock KG, Todd C, Wareham K. Investigating the feasibility of recruitment to an observational, quality-of-life study of patients diagnosed with atrial fibrillation (AF) who have experienced a bleed while anticoagulated: EQUAL-AF feasibility study protocol. Pilot Feasibility Stud. 2022 Aug 12;8(1):180. doi: 10.1186/s40814-022-01135-8. PMID 35962446
- See also: Related Info — http://hbr.org/2013/10/the-strategy-that-will-fix-health-care

DOCUMENTS (1):
  • Study Protocol (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04921176/Prot_000.pdf